CLINICAL TRIAL: NCT04180241
Title: Development of Endoscopic Treatment for Achalasia, POEM (Per Oral Esophageal Myotomy): A Randomized Controlled Trial
Brief Title: Development of Endoscopic Treatment for Achalasia
Acronym: POEM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anders Thorell, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017/1630-31
Record Dates: First submitted 2019-11-07; First posted 2019-11-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Intervention Model Description: POEM with division all the esophageal muscle layers compared to deviding only the inner circular muscle layer of the esophagus.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization process is initiated after general anesthesia is induced and the group affiliation will be determined by opening of a sealed envelope specifying the group assignment. The information of group allocation is stored in a closed envelope kept in a locked archive until the study is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- total division of the muscle layer (Active Comparator): POEM- total division of the circular muscle layer into the gastroesophageal junction
  Interventions: Procedure: POEM
- partial division of the muscle layer (Active Comparator): POEM - partial division of the circular muscle layer into the gastroesophageal junction
  Interventions: Procedure: POEM

INTERVENTIONS:
Procedure: POEM — Peroral endoscopic myotomy

SUMMARY:
Per Oral Endoscopic Myotomy (POEM); comparison of two surgical techniques division all the esophageal muscle layers versus division the inner circular muscle layer of the esophagus only.

DETAILED DESCRIPTION:
Prior to surgery, all patients undergo upper endoscopy , x-ray "time barium" manometry, 24 hours pH registration. Moreover Quality of Life instrument (RAND-36), GSRS (Gastrointestinal Symptom Rating Scale) and a dysphagia score (Eckardt score) are completed by all patients.

Follow-up with surveys 3, 6, 12, and 36 months (GSRS, RAND-36 and Eckardt score).

At 3,12 and 36 months an x-ray "time barium" is performed and after 12 months a gastroscopy and at 24 hours esophageal pH monitoring are performed.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed achalasia
* the patient should understand the nature and the purpose of the study and give informed consent

Exclusion Criteria:

* previous surgical treatment of achalasia
* inability to understand the contents of or follow the protocol
* other pathology as an explanation for the obstruction of the esophageal transition

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who develop gastroesophageal reflux disease (GERD) | 1 year
  Measured as esophageal acid exposure (pH <4) > 4% of recorded time

SECONDARY OUTCOMES:
Esophageal emptying function | 1 year
  Measured by Time Barium Swallow X-ray
Eckardt score | 1 year
  The Eckardt score consists of 4 components including dysphagia, chest pain, regurgitation, and weight loss.Each component is assigned a score from 0 to 3 based on the patient's self-reported response, resulting in a total score that can vary from 0 to 12, higher scores mean a worse outcome.
RAND-36 | 1 year
  The RAND-36 It is comprised of 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions. Physical and mental health summary scores are also derived from the eight RAND-36 scales. higher scores mean a better outcome.
Dysmotility | 1 year
  measured by Manometry
Gastrointestinal Symptom Rating Scale (GSRS) | 1 year
  Scoring;The questionnaire, which contains 15 items, uses a seven-graded Likert scale, where 1 represents the most positive option and 7 the most negative one.
  A mean value for the items in each dimension should be calculated:
  Diarrhoea syndrome: 11. Increased passage of stools 12. Loose stools 14. Urgent need for defecation Indigestion syndrome: 6. Borborygmus 7. Abdominal distension 8. Eructation 9. Increased flatus Constipation syndrome: 10. Decreased passage of stools 13. Hard stools 15. Feeling of incomplete evacuation Abdominal pain syndrome: 1. Abdominal pain 4. Sucking sensations 5. Nausea and vomiting Reflux syndrome: 2. Heartburn 3. Acid regurgitation

CONTACTS AND LOCATIONS:
Overall Officials: Anders Thorell, Professor, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Karolinska Institutet, Ersta Hospital, Stockholm, Region Stockholm
  - Karolinska Institutet, Stockholm, Stockholm County Council